CLINICAL TRIAL: NCT02301585
Title: Optimization of Fluid Therapy by a Passive Leg Raising Test in Patients With Septic Shock in the ICU
Brief Title: Optimization of Fluid Therapy in Sepsis by a Passive Leg Raising Test
Acronym: OFTaPLR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because of futility due to unexpected low weight gain in both groups.
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Svenska militärläkarföreningen (Unknown)
Responsible Party: Principal Investigator, Christer Svensen, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLR EPN 2013/1337-31/2
Record Dates: First submitted 2014-09-14; First posted 2014-11-26 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Shock, Septic
Keywords: shock, septic; hemodynamics; algorithms
MeSH Terms: conditions — Shock, Septic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passive Leg Raising (Experimental): Before decision on fluid administration a passive leg raising test is performed. If the test indicates fluid irresponsiveness optimization of circulation will be done with vasopressors or inotropes.
  Interventions: Procedure: Passive Leg Raising Test
- Standard of care (Active Comparator): Patients are treated according to Surviving Sepsis Guidelines. Fluid is administered according to the choice of the clinician.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Passive Leg Raising Test — Before decision on fluid administration a passive leg raising test is performed. The results are interpreted according to a treatment protocol. If the test indicates fluid irresponsiveness optimization of circulation will be done with vasopressors or inotropes.
  Arms: Passive Leg Raising
Procedure: Standard of care — Patients are treated according to Surviving Sepsis Guidelines
  Arms: Standard of care

SUMMARY:
A randomized controlled clinical trial to evaluate whether a passive leg raising test to guide fluid therapy of patients with septic shock can reduce fluid balance and weight gain. Patients will be treated according to an algorithm in which the indexed stroke volume (stroke volume related to body surface area) and mean arterial pressure will guide the timing and amount of fluid and the use of inotropic and vasoactive support. Patients will be randomized to either an intervention group in which a passive leg raising test will be made prior to any decision for fluid administration or to a control group where this test is not performed and fluid administration is carried out according to standard of care at the department.

Hypothesis: A passive leg raising test, will reduce weight gain by day 3 by 30%.

ELIGIBILITY:
Inclusion Criteria:

All patients >18 years admitted to the ICU diagnosed with circulatory shock due to suspected sepsis or pancreatitis. Circulatory shock is defined as MAP<70 mm Hg or need for norepinephrine despite resuscitation with ≥30 ml/kg of crystalloid fluids.

Exclusion Criteria:

> 12 hours have passed after onset of shock. The patient has contraindications for an arterial femoral/axillary line. Elevated ICP. Patients who have had a femoral amputation. Elevated intraabdominal pressure>20 cm H2O.

Suspension criteria: The patient has developed pulmonary oedema during PLR test. Life threatening bleeding.

Serious adverse events:

Trombosis in arteria femoralis. Death during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
weight gain | 3 days

SECONDARY OUTCOMES:
ICU length of stay | measured within 90 days after inclusion
  Number of days spent in the ICU: time and date of discharge from the ICU minus time and date of admission to the ICU. A started but not yet completed day is counted as one.
Cumulative fluid balance study day 1,2,3 | Study day 1,2,3
  Fluids in-Fluids out during the study period.
30 day mortality | 30 days from inclusion in the study
  Is the patient alive or dead after 30 days?
Organ support during ICU stay | ICU-stay
  Number of days with mechanical ventilation, vasopressors/inotropic support, CRRT.
ICU discharge status | End of ICU stay
  Alive or dead at discharge from the ICU?

CONTACTS AND LOCATIONS:
Overall Officials: Christer Svensen, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Södersjukhuset, Stockholm, Sweden